CLINICAL TRIAL: NCT02135783
Title: A Randomised Trial to Establish the Efficacy and Safety of Decompressive Craniectomy Combined With Hematoma Removal in Patients With Intracerebral Hemorrhage
Brief Title: Decompressive Craniectomy Combined With Hematoma Removal to Treat ICH
Acronym: CARICH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Rong Hu, Associate Professor, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Neurosurg 01
Record Dates: First submitted 2014-05-07; First posted 2014-05-12 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Intracranial Hemorrhages
MeSH Terms: conditions — Intracranial Hemorrhages | interventions — Decompressive Craniectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Decompressive Craniectomy (Experimental): Decompressive Craniectomy afte Hematoma Removal in Patients with Intracerebral Hemorrhage
  Interventions: Procedure: Decompressive Craniectomy
- non-Decompressive Craniectomy (Active Comparator): non-Decompressive Craniectomy afte Hematoma Removal in Patients with Intracerebral Hemorrhage
  Interventions: Procedure: non-Decompressive Craniectomy

INTERVENTIONS:
Procedure: Decompressive Craniectomy — A portion of frontal,temporal, and parietal bone was removed by craniectomy and the size of decompression was about 10x12 cm2.Intracerebral hematoma was evacuated by transcortical approach with the aid of a surgical microscope.
  Arms: Decompressive Craniectomy
Procedure: non-Decompressive Craniectomy — a simple hematoma removal by osteoplastic craniotomy group (HR) or Intracerebral hematoma was evacuated by transcortical approach with the aid of a surgical neuroendoscopyand the size of decompression was about 3x2.5 cm2.
  Arms: non-Decompressive Craniectomy

SUMMARY:
Decompressive craniectomy has been reported for the treatment of patients with intracerebral hemorrhage. But no prospective randomised controlled trials have yet been undertaken to confirm its effect.The purpose of the study is to determine whether decompressive craniectomy post hematoma removal surgery after intracerebral hemorrhage will reduce the chances of a person dying or surviving with a long term disability.

DETAILED DESCRIPTION:
Intracerebral hemorrhage (ICH) is one of the most serious subtypes of stroke, affecting approximately 2-3 million people worldwide each year. About one third of people with ICH die early after onset and the majority of survivors are left with major long-term disability. Hematoma removal (HR) surgery is the primary treatment for ICH which volume is more than 30ml. But whether decompressive craniectomy (DC) should be employed during the HR surgery still has considerable controversy. Outcomes in this study will be measured at 3 months after surgery via a postal questionnaire including the Glasgow Outcome scale, Modified Rankin Scale, and Barthel index. Two hundred patients will be recruited to the trial over 36 months. Follow-up will take three months with analysis and reporting taking one year.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a spontaneous lobar and basal ganglia ICH on CT scan
* Patient within 72 hours of ictus
* Best score on the GCS of 5-13.
* Volume of hematoma between 30 and 100ml [Calculated using (a x b x c)/2 method]
* The history of hypertensive

Exclusion Criteria:

* Clear evidence that the hemorrhage is due to an aneurysm or angiographically proven arteriovenous malformation.
* Intraventricular hemorrhage of any sort
* ICH secondary to tumour or trauma.
* If the hematological effects of any previous anticoagulants are not completely reversed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Mortality and disability | 3 months
  according to a 3-6 scores on the modified Rankin Score

SECONDARY OUTCOMES:
Occurrence of second Surgery | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rong Hu, MD,PhD, Principal Investigator — Department of Neurosurgery, Southwest Hospital
Locations (1):
- Department of Neurosurgery , Southwest Hospital, Third Military Medical University,, Chongqing, China

REFERENCES:
- [Derived] Zhang C, Zhang S, Yin Y, Wang L, Li L, Lan C, Shi J, Jiang Z, Ge H, Li X, Ao Z, Hu S, Chen J, Feng H, Hu R. Clot removAl with or without decompRessive craniectomy under ICP monitoring for supratentorial IntraCerebral Hemorrhage (CARICH): a randomized controlled trial. Int J Surg. 2024 Aug 1;110(8):4804-4809. doi: 10.1097/JS9.0000000000001466. PMID 38640513
- [Derived] Hu R, Zhang C, Xia J, Ge H, Zhong J, Fang X, Zou Y, Lan C, Li L, Feng H. Long-term Outcomes and Risk Factors Related to Hydrocephalus After Intracerebral Hemorrhage. Transl Stroke Res. 2021 Feb;12(1):31-38. doi: 10.1007/s12975-020-00823-y. Epub 2020 Jun 8. PMID 32514905